CLINICAL TRIAL: NCT06607029
Title: Opioid-free Anesthesia Protocol on the Quality of Recovery After Neurosurgical Supratentorial Tumor Resection: A Randomized, Controlled, Clinical Trial
Brief Title: Opioid-free Anesthesia Protocol for Neurosurgical Supratentorial Tumor Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Ruquan Han, Head of Anesthesiology, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OFA20240914
Record Dates: First submitted 2024-09-15; First posted 2024-09-23 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-03

CONDITIONS: Supratentorial Tumors
MeSH Terms: conditions — Supratentorial Neoplasms

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the opioid-based control group (Active Comparator)
  Interventions: Drug: the opioid-based control group
- the opioid-free anaesthesia group (Experimental)
  Interventions: Drug: the opioid-free anesthesia group

INTERVENTIONS:
Drug: the opioid-based control group — Intraoperative analgesia will be administered with conventional opioid drugs such as sufentanil and remifentanil.
  Arms: the opioid-based control group
Drug: the opioid-free anesthesia group — The patients will be administered with an opioid-free strategy during surgery. The investigator will use esketamine, dexmetopidine, and local anesthesia to control perioperative pain.
  Arms: the opioid-free anaesthesia group

SUMMARY:
Opioids have many side effects, such as constipation, urinary retention, itchy skin, respiratory depression, and postoperative nausea and vomiting. These side effects can lead to delayed recovery, longer hospital stays, and increased health care costs. Opioid-free anesthesia is the combination of anti-nociceptive drugs to block the different pathways involved in the transmission of nociceptive information, control pain, avoid opioid-related adverse reactions, and promote patient recovery. At present, opioid-free anesthesia is not widely used in craniocerebral surgery in neurosurgery, and the relevant clinical data are extensive. Therefore, the investigators urgently need to conduct a randomized controlled study to provide clinical evidence for the efficacy and safety of opioid-free anesthesia in neurosurgical patients.

DETAILED DESCRIPTION:
Data sharing plan: The deidentified participant data reported in this study could be made available to researchers upon approval by the corresponding author (Dr. Ruquan Han, ruquan.han@ccmu.edu.cn) immediately after publication. The reasonable request should provide a formal protocol for database use that has been approved by the ethics institutions.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled to undergo craniotomy for supratentorial tumors with general anesthesia;
* 18 years≤age≤65 years;
* American Society of Anesthesiologists (ASA) physical status of I to III;
* Signed informed consent.

Exclusion Criteria:

* Patients with a body mass index (BMI)≥35 kg/m2;
* Patients with severe hepatic and renal insufficiency;
* Patients with cognitive dysfunction, aphasia and other states that do not cooperate with the assessment;
* Preoperative magnetic resonance imaging of the head showed midline displacement >5 mm;
* Patients undergoing electrophysiological monitoring during surgery;
* Pregnant or lactating patients.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 170 (Estimated)
Dates: Start 2024-10-21 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
the quality of recovery-15(QoR-15) score on the second day after surgery | on the second day after surgery
  Quality of Recovery-15(QoR-15) score, as a tool to evaluate recovery quality during perioperative period. The QoR-15 scale was used to assess patients' postoperative recovery. Each item is scored on a 10-point scale, from 0 (worst recovery) to 150 (best recovery).

SECONDARY OUTCOMES:
The QoR-15 score on the 5th day after surgery | on the 5th day after surgery
The incidence of nausea and vomiting within 48 hours after surgery | 48 hours after surgery
The NRS pain score on the second and 5th days after surgery | on the second and 5th days after surgery
The sleep quality on the second and 5th days after surgery | on the second and 5th days after surgery
The incidence of chronic pain at 3 and 6 months after surgery | at 3 and 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Yes
Data sharing plan: The deidentified participant data reported in this study could be made available to researchers upon approval by the corresponding author (Dr. Ruquan Han, ruquan.han@ccmu.edu.cn) immediately after publication. The reasonable request should provide a formal protocol for database use that has been approved by the ethics institutions.

REFERENCES:
- [Derived] Fu Y, Zhou Y, Cui Y, Wu Y, Wang T, Li Y, Yu Y, Han R. Opioid-free anaesthesia and postoperative quality of recovery in patients undergoing supratentorial tumour resection: protocol for a randomised controlled trial. BMJ Open. 2025 May 15;15(5):e099864. doi: 10.1136/bmjopen-2025-099864. PMID 40379317